CLINICAL TRIAL: NCT02214290
Title: Effect of Oral Caffeine and L-Citrulline Supplementation on Arterial Function in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HSC2013.10514
Record Dates: First submitted 2014-08-04; First posted 2014-08-12 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-10

CONDITIONS: Hypertension; Healthy
Keywords: Cardiovascular; Caffeine; L-citrulline; Arterial Function; Hemodynamics; Blood Pressure; Pulse Wave Velocity; Pulse Wave Analysis
MeSH Terms: conditions — Hypertension | interventions — Caffeine; Citrulline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Caffeine (Active Comparator): 200 mg caffeine tablet produced by CVS Pharmacy, USA
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Placebo pill produced by NOW FOODS, USA
  Interventions: Drug: Placebo
- L-citrulline (Experimental): L-citrulline capsule (750 mg) provided by NOW FOODS
  Interventions: Dietary Supplement: L-citrulline

INTERVENTIONS:
Drug: Caffeine — A 200 mg caffeine tablet was given to subject to examine the drugs effect on arterial function.
  Other Names: Caffeine tablet (CVS Pharmacy)
  Arms: Caffeine
Drug: Placebo — A 750 mg placebo capsule (maltodextrin) was given to subjects to examine the effect of the drug on arterial function.
  Other Names: Placebo from NOW FOODS, USA
  Arms: Placebo
Dietary Supplement: L-citrulline — L-citrulline was used to examine the effect of the supplement on arterial function.
  Other Names: L-citrulline (750 mg/capsule)
  Arms: L-citrulline

SUMMARY:
Caffeine is an exceedingly popular and consumed pharmacological agent. Although caffeine is primarily consumed from coffee and tea beverages, it is also available in other forms such as sodas, energy drinks, tablets and capsules. Nevertheless, caffeine acutely increases brachial and aortic systolic blood pressure (BP) and arterial stiffness. Arterial stiffness is an independent predictor of cardiovascular disease (CVD) and assessed through pulse wave velocity (PWV). Interestingly, previous studies have proposed that caffeine may increase aortic BP through increases in aortic PWV and augmentation index (AIx), a measurement of wave reflection. Yet, these effects were seen in middle-aged adults with treated hypertension and a wide age range. Therefore, it is imperative to consider that caffeine may cause different effects in young normotensive individuals than in older adults independently of BP levels. Importantly, oral supplementation of the amino-acid, L-citrulline has been shown to enhance the bioavailability of L-arginine levels and nitric oxide (NO) production and, therefore, improve arterial function. L-citrulline supplementation for 7 days given at 6 g/day has shown to increase NO levels while improving PWV. Previous studies by our group also demonstrated that L-citrulline supplementation reduces the BP response to cold exposure; a condition with an increased vasoconstriction. Therefore, the acute effects of caffeine on central and peripheral PWV and BP in healthy young men are yet to be fully evaluated. We hypothesized that acute caffeine intake would increase peripheral and aortic BP and PWV and that L-citrulline supplementation would attenuate the effects induced by acute caffeine ingestion.

DETAILED DESCRIPTION:
The specific aims of this study are:

AIM 1: To examine the effects of the acute ingestion of 200mg caffeine (tablets) on arterial function in young adults. The working hypothesis is that acute caffeine intake would increase brachial, ankle and aortic BP, PWV (aortic and leg), and wave reflection. In order to test this hypothesis, the investigators will perform non-invasive measurements of arterial stiffness (aortic and leg PWV) and pulse wave analysis (aortic BP and AIx) using applanation tonometry of the radial artery 30, 45, and 60 minutes following caffeine ingestion.

AIM 2: To determine the effectiveness of L-citrulline supplementation to attenuate the acute cardiovascular effects of caffeine ingestion. The working hypothesis is that 7 days of L-citrulline supplementation will attenuate the unfavorable arterial responses (increases in BP, PWV, and wave reflection) to acute caffeine ingestion. In order to test this hypothesis, the investigators will perform the same procedures previously specified in AIM 1.

Description of the study:

Sixteen healthy young men 18-40 years of age will be enrolled in this study. Participants with CVD history, resting BP (> 160/100 mmHg), recent history of smoking, or considered competitive athlete will be excluded from the study. All subjects will refrain from food and caffeine for > 8 hours and from exercise for > 24 hours before testing.

Study design:

Following an initial screening, arterial function measurements will be collected. Measurements will be assessed at baseline following 10 minutes of rest in the supine position and then again at 30, 45, and 60 minutes after 200 mg caffeine or placebo ingestion. Participants will receive caffeine or placebo supplementation on two separate visits with a minimum of 48 hours in between sessions. Following the acute phase of the study, subjects will be randomized to consume L-citrulline or placebo for 7 days given at 6 grams/day. Following the same protocol as the acute phase with 200 mg caffeine, measurements will be collected before and after the 7 day supplementation period.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy males
* Non smoker
* Non endurance trained athlete
* No previous history of cardiovascular disease

Exclusion Criteria:

* Female
* Blood pressure greater than 160/100
* Smoker

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, M.D. Ph.D, Principal Investigator — Florida State University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen young healthy men participated in this study. All subjects were non-smokers, recreationally active, and free of apparent cardiovascular-metabolic diseases based on medical history.
Pre-assignment Details: Of the 42 individuals screened, 16 individuals completed the intervention in its entirety.
Groups:
- Citrulline First, Then Placebo: Each participant received L-Citrulline (6g/day) for a 7 day period. This was followed by a 14 day washout period. Finally, the same participants then received a Placebo (6g/day maltodextrin) for a 7 day period.
- Placebo First, Then L-Citrulline: Each participant received a Placebo (6g/day maltodextrin) for a 7 day period. This was followed by a 14 day washout period. Finally, the same participants then received a L-Citrulline (6g/day) for a 7 day period.
Period: First Intervention (7 Days)
Arm/Group | Citrulline First, Then Placebo | Placebo First, Then L-Citrulline
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Citrulline First, Then Placebo | Placebo First, Then L-Citrulline
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Citrulline First, Then Placebo | Placebo First, Then L-Citrulline
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- L-Citrulline or Placebo: Placebo and L-Citrulline pills produced by NOW FOODS, USA
  Citrulline or Placebo (both 6g/day) were given for a 7 day supplementation period. This was followed by a 14 day washout period and crossover to the other supplement (L-Citrulline or Placebo) for 7 days. Measurements of arterial function were performed to determine if the supplements had any significant effect on blood pressure control/pressure wave reflection at rest and immediately after ingestion of 200 milligrams of caffeine.
Arm/Group | L-Citrulline or Placebo
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — ages of 18 to 40 years
  years | 23 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Aortic Blood Pressure
Description: Aortic blood pressure at rest and 30 minutes after acute ingestion of 200 mg of caffeine before and after 7 days of either 6g/day of Citrulline or 6 g/day of Placebo.
Time Frame: Baseline and Day 7 (Calculated change between rest and 30 minutes post-caffeine ingestion at these time points)
Population: Young, apparently healthy individuals, aged 18-40 years old.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Citrulline: Participants received 6g/day of Citrulline for 7 days
- Placebo: Participants received 6 g/day of Maltodextrin for 7 days.
Arm/Group | Citrulline | Placebo
Number analyzed (Participants) | 16 | 16
mmHg
  Baseline | 5 (1) | 6 (1)
  7 Days | 4 (1) | 4 (1)
Statistical Analysis 1: Comparison: Citrulline vs Placebo; Test type: Other; p < 0.001, ANOVA; post-hoc comparisons were used to determine within-group and between-group differences

2. Secondary Outcome: Changes in Reflected Wave Pressure (P2)
Description: Reflected wave pressure at rest and 30 minutes after ingestion of 200mg of caffeine after 7 days supplementation of 6g/day of either L-Citrulline or Placebo.
Time Frame: Baseline and Day 7 (Calculated change between rest and 30 minutes post-caffeine ingestion at these time points)
Population: Young, apparently healthy adults, aged 18-40 years.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Participants received 6 g/day of Placebo
Arm/Group | Citrulline | Placebo
Number analyzed (Participants) | 16 | 16
mmHg
  Baseline | 5 (1) | 5 (1)
  7 Days | 4 (1) | 5 (1)
Statistical Analysis 1: Comparison: Citrulline vs Placebo; Test type: Other; p < 0.001, ANOVA; post-hoc comparisons were used to determine within-group and between-group differences

3. Secondary Outcome: Changes in Femoral-ankle Pulse Wave Velocity After 7 Days of Either L-Citrulline or Placebo (6g/Day)
Description: Femoral-ankle pulse wave velocity at rest and 30 minutes after ingestion of 200mg of caffeine after 7 days supplementation of 6g/day of either L-Citrulline or Placebo.
Time Frame: Baseline and Day 7 (Calculated change between rest and 30 minutes post-caffeine ingestion at these time points)
Population: young, apparently healthy adults, aged 18-40 years
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Citrulline: Participants received a 6 g/day of Citrulline for 7 days
- Placebo: Participants received a 200 mg maltodextrin tablet, and femoral-ankle pulse wave velocity was taken at 60 minutes post-ingestion.
Arm/Group | Citrulline | Placebo
Number analyzed (Participants) | 16 | 16
m/s
  Baseline | 0.6 (0.4) | 0.7 (0.5)
  7 Days | 0.4 (0.4) | 0.6 (0.4)
Statistical Analysis 1: Comparison: Citrulline vs Placebo; Test type: Other; p < 0.001, ANOVA; post-hoc comparisons were used to determine within-group and between-group differences

ADVERSE EVENTS:
Description: Adverse events were not monitored/assessed because the participants were young and healthy.
Groups:
- Placebo: Participants received 6g/day of Placebo (Maltodextrin) for 7 days
Arm/Group | Citrulline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No